CLINICAL TRIAL: NCT02285309
Title: The Utility of Novel Measurements of Diastolic Function Involving Transoesophageal and Transthoracic Echocardiography in the Peri-operative Period in Patients Undergoing Cardiac Surgery -an Exploratory Trial
Brief Title: Perioperative Measurements of Diastolic Function in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: UCLondon
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Diastolic Dysfunction
Keywords: Cardiac Surgery; Diastolic Dysfunction; Enoximone
MeSH Terms: interventions — Cardiac Surgical Procedures; Enoximone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac surgery
  Interventions: Procedure: Cardiac Surgery and enoximone

INTERVENTIONS:
Procedure: Cardiac Surgery and enoximone — Does diastolic function change with cardiac surgery +/- enoximone

SUMMARY:
This observational clinical trial will investigate the following perioperative indices relating to cardiac surgery:

1. The significance of measurements involving left heart relaxation (LV diastolic function) and its relation to outcome measures.
2. The significance of measurements involving right heart relaxation function and itrs relation to outcome measures.
3. The influence of drugs such as enoximone on these outcome measures.

DETAILED DESCRIPTION:
Over the past two decades, perioperative TOE has become routine part of monitoring in the setting of cardiac surgery. In many centres around the world nearly 100% of pateints undergoing cardiac surgery are monitored using this modality. There are several studies and observational reviews suggesting intraoperative TOE can change management and thus indirectly influence outcome in patients undergoing valve, aortic or bypass graft surgery. Certainly in our centre at The Heart Hospital, it is routine practce to perform an intraoperative TOE in all patients undergoing cardiac surgery in order to guide surgical and anaesthetic management of the patient. Despite this use of TOE there is very little evidence of how TOE influences patient related outcomes, both morbidity and mortality.

Several advances have occurred over the years involving both better technology to image the heart with TOE along with the development of novel measurements of heart function. As technology has evolved, many modalities and measurement have not been validated in the setting of cardiac surgery. In our observational clincal trial we aim to investigate the following:

1. The significance of measurements involving left heart relaxation (LV diastolic function) and its relation to outcome measures.
2. The significance of measurements involving the right heart relaxation function and itrs relation to outcome measures.
3. The influence of drugs such as enoximone on these outcome measures.

While many of these measurements have been validated in the care of medical patients, they have not been examined in the surgical setting. In addition, its ability to predict outcome has never been tested. We believe this study will help us answer these important questions.

ELIGIBILITY:
Inclusion Criteria:

* Systolic dysfunction (EF <50%) or diastolic dysfunction grade 1-3 as determined through preoperative TTE or intraoperative TOE
* Able to give informed consent

Exclusion Criteria:

* Contraindication to transoesphageal echocardiography (such as previous oesophagectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change in diastolic dysfunction -categorised as improved, stable or worse | Up to 12 hours
  Compare diastolic dysfunction before and after surgery in those that receive enoximone. Compare diastolic function before and after surgery in those that do not receive enoximone

SECONDARY OUTCOMES:
Systolic and diastolic data from the post operative transthoracic echocardiogram | Up to 30 days
  Compare systolic and diastolic function on transthoracic echocardiography to intraoperative parameters
Duration of endotracheal intubation (in hours) | 0-30 days
  How long patient remains intubated on ICU post operatively
Incidence of post operative atrial fibrillation | 0-30 days
  As above
Duration of ICU stay | 0-30 days
  As above
Duration of hospital stay | 0-30 days
  As above
Cardiac Post Operatie Morbidity Score (C-POMS) | 0-30 days
  As above
30 day Major Adverse Cardiovascular Events | 0-30 days
  As above